CLINICAL TRIAL: NCT06715904
Title: Comparison of the Effect of a Morton's Extension on Plantar Pressure Distribution in Different Foot Regions in Female and Male Patients Without Deformities: A Pre-Post Test Study
Brief Title: Sex Differences in Morton's Extension Application on Plantar Pressure Distribution in Different Foot Regions in Female and Male Patients Without Deformities: A Pre-Post Test Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist., Mayuben Private Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/235(B)-E
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: metatarsalgia; Foot; orthopedics; women
MeSH Terms: conditions — Metatarsalgia | interventions — Orthopedic Procedures

STUDY DESIGN:
Intervention Model Description: Sex research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women (Experimental): A Morton extension with a height of 5 mm was insert from the proximal area of the first metatarsal head to the base of the proximal phalanx of the Hallux.
  Interventions: Other: Womens with Morton´s Extension
- Men (Experimental): A Morton extension with a height of 5 mm was insert from the proximal area of the first metatarsal head to the base of the proximal phalanx of the Hallux.
  Interventions: Other: Womens with Morton´s Extension

INTERVENTIONS:
Other: Womens with Morton´s Extension — Morton extension application
  Other Names: Orthopaedics

SUMMARY:
The aim of this study is to simulate the orthopedic treatment called Morton's extension on non-deformed patients to check the different effects producted by sex in footprint.

DETAILED DESCRIPTION:
The objective of this study is to perform an assimilation of the orthopedic treatment called morton extension on non-deformed patients to verify the difference effects due by sex on each metatarsal head and rearfoot on its static footprint, and plantar pressures variables in dynamic footprint.

ELIGIBILITY:
Inclusion Criteria:

* no history of trauma to the foot;
* the presence of at least 10° of dorsiflexion at the ankle with the knee fully dorsiflexed;
* unrestricted motion of the functional subtalar joint of 30°;
* unrestricted motion along the longitudinal axis of the midtarsal joint of 15°;
* unrestricted nonweight-bearing motion of the first ray of at least 8 mm;
* greater than 50° of dorsiflexion of the hallux to the first metatarsal bisection during nonweight-bearing;
* age greater than 18 years and younger than 60 years;
* at the time of data collection, no lower limb dysfunction or chronic injury; and
* no evidence of a non-fixed deformity at first metatarsophalangeal and first metatarsal cuneiform joints.

Exclusion Criteria:

* plantar corns and calluses,
* hallux valgus and lesser toe deformities,
* diabetes,
* any abnormality in the lower extremity that may affect gait.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — comparative study by sex of Morton´s extension effects
Enrollment: 50 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Before Morton Extension Medium pressure | Through study completion, an average of 1 week.
  Static footprint will measure medium plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
Extension Maximum pressure | Through study completion, an average of 1 week.
  Static footprint will measure maximum plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
After Morton Extension Medium pressure | Through study completion, an average of 1 week.
  Static footprint will measure medium plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
After Morton Extension Maximum pressure | Through study completion, an average of 1 week
  Static footprint will measure maximum plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
Before Morton Extension Medium pressure | Through study completion, an average of 1 week
  Dynamic footprint will measure medium plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
Before Morton Extension Maximum pressure | Through study completion, an average of 1 week
  Dynamic footprint will measure maximum plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
After Morton Extension Medium pressure | Through study completion, an average of 1 week
  Dynamic footprint will measure medium plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
After Morton Extension Maximum pressure | Through study completion, an average of 1 week
  Dynamic footprint will measure maximum plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Sanchez-Serena, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No